CLINICAL TRIAL: NCT05922150
Title: Efficiency of Low Level Laser Therapy and Ozone on Sequelae After Extraction of Impacted Mandibular Third Molar
Brief Title: Effect of LLLT and Ozone to Reduce Complications After Extraction of Impacted Lower Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Osama Abdulkathim Ali, postgraduate student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LLLT & ozone
Record Dates: First submitted 2023-05-27; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Complications of Extraction of Impacted Teeth
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LLLT and ozone group (Experimental): administered of low level laser therapy and ozone gel after extraction of impacted mandibular third molar
  Interventions: Radiation: low level laser therapy; Drug: ozone gel
- LLLT group (Experimental): administered of low level laser therapy after extraction of impacted mandibular third molar
  Interventions: Radiation: low level laser therapy
- ozone group (Experimental): administered of low ozone gel after extraction of impacted mandibular third molar
  Interventions: Drug: ozone gel
- control group (No Intervention): routinely extraction of impacted mandibular third molar

INTERVENTIONS:
Radiation: low level laser therapy — LLLT induces cellular biostimulation, speeds up tissue regeneration, enhances wound healing, and reduces pain and swelling through an anti-inflammatory effect. This is because the LLLT increases phagocytic activity, and the number and diameter of lymphatic vessels, decreases the permeability of blood vessels and restores microcapillary function
  Arms: LLLT and ozone group; LLLT group
Drug: ozone gel — ozone is effective antimicrobial (viricidal, bactericidal, and fungicidal). Other well-known benefits include immunological modulatory and stimulating effects and anti-inflammatory, biosynthetic, anti-hypoxic, and bioenergeticseffects
  Arms: LLLT and ozone group; ozone group

SUMMARY:
Many factors cause third molars to stay impacted in the jaws, hence the extraction of impacted wisdom teeth occurs often in dental clinics. Pain, trismus, and edema are typical postoperative complications following third molar surgery. Various strategies have been developed to prevent or reduce these postoperative complications, Among these is the use of Low-Level Laser Therapy (LLLT), which demonstrates numerous benefits in lowering pain, trismus, and edema by managing inflammation. The precise biological mechanism of action remains unknown. There seems to be evidence that it may have neuro-pharmacological impacts on the production, metabolism, and release of a number of biological compounds, the other option is use of ozone which has antimicrobial effectiveness (viricidal, bactericidal, and fungicidal). Additional well-known advantages include immunological modulatory and stimulating actions, including anti-inflammatory, biosynthetic, anti-hypoxic, and bioenergetic characteristics. Ozone can interact with blood components in the right amounts to positively impact oxygen metabolism and cell energy while also triggering antioxidant defense mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Patients who had mandibular third molar, totally or partially impacted in the bone (Class II-III and position B, Pell and Gregory's classification), in need of surgical extraction, which were evaluated clinically and by radiological examination.
* Patients who were in age range between 18-40 years old.
* Patients who were willing to compliance with study and were available for follow up.
* Patients should be with good oral hygiene and without any acute illness

Exclusion Criteria:

* Patients with medical condition that prevent any surgical intervention such as patient with recent myocardial infarction, bleeding disorders, psychiatric problem and patients with pacemaker, uncontrolled systemic disease, immunocompromised patient and patients taking corticosteroid and anti-inflammatory drugs.
* Patients with history of head and neck radiotherapy.
* Pregnant or lactation women
* Active advanced uncontrolled periodontal disease and bad oral hygiene, or patients with local acute infection in relation to third molar especially pericoronitis.
* Patients who suffer from photodermatoses and photosensitized patients (photoallergies).
* Hyperthyroidism

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
pain | baseline to seventh day
  measurement of pain by NRS, between 0 and 10, zero meaning no pain and 10 meaning worst imaginable pain
swelling | baseline to seventh day
  measurement of swelling by using tape, using 3 lines
trismus | baseline to seventh day
  measurement of maximum mouth opening by using digital Vernia

CONTACTS AND LOCATIONS:
Locations (1):
- Osama, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Result] Eshghpour M, Ahrari F, Takallu M. Is Low-Level Laser Therapy Effective in the Management of Pain and Swelling After Mandibular Third Molar Surgery? J Oral Maxillofac Surg. 2016 Jul;74(7):1322.e1-8. doi: 10.1016/j.joms.2016.02.030. Epub 2016 Mar 12. PMID 27055228
- [Result] Roynesdal AK, Bjornland T, Barkvoll P, Haanaes HR. The effect of soft-laser application on postoperative pain and swelling. A double-blind, crossover study. Int J Oral Maxillofac Surg. 1993 Aug;22(4):242-5. doi: 10.1016/s0901-5027(05)80646-0. PMID 8409569
- [Result] Kazancioglu HO, Ezirganli S, Demirtas N. Comparison of the influence of ozone and laser therapies on pain, swelling, and trismus following impacted third-molar surgery. Lasers Med Sci. 2014 Jul;29(4):1313-9. doi: 10.1007/s10103-013-1300-y. Epub 2013 Mar 14. PMID 23494104